CLINICAL TRIAL: NCT00258817
Title: Annual Study for Serum Collection and Evaluation of Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Influenza Virus Vaccine (2005-2006 Formulation)
Brief Title: Phase IV Trial to Collect Safety Data and Sera in Healthy Children Given Fluzone Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC26
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Results first posted 2009-03-25 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Fluzone®; Influenza Virus Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza Virus Vaccine Naïve (Experimental): Subjects have never received Influenza virus vaccine in the past
  Interventions: Biological: Influenza Virus Vaccine (Fluzone®)
- Influenza Virus Vaccine-primed (Experimental): Subjects have received Influenza virus vaccine in the past
  Interventions: Biological: Influenza Virus Vaccine (Fluzone®)

INTERVENTIONS:
Biological: Influenza Virus Vaccine (Fluzone®) — 0.25 mL, Intramuscular (Day 0 and Day 28)
  Other Names: Fluzone®
  Arms: Influenza Virus Vaccine Naïve
Biological: Influenza Virus Vaccine (Fluzone®) — 0.25 mL, Intramuscular (Day 0)
  Other Names: Fluzone®
  Arms: Influenza Virus Vaccine-primed

SUMMARY:
To provide serum to the Food and Drug Administration (FDA) for use by FDA, the Centers for Disease Control and Prevention (CDC), and the World Health Organization (WHO) for characterization of circulating influenza strains.

Observational Objectives:

To describe the safety of the 2005-2006 pediatric formulation of Fluzone vaccine, given in the two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to < 36 months.

To describe the immunogenicity of the 2005-2006 pediatric formulation of Fluzone vaccine, administered in a two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to < 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged ≥ 6 months (24 weeks) to < 36 months (3rd birthday).
* Participant is considered to be in good health on the basis of reported medical history and limited physical examination.
* Participant is available for the duration of the study.
* Parent/legal acceptable representative is willing and able to provide informed consent.
* Parent/legal acceptable representative is willing and able to meet protocol requirements.
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg.

Exclusion Criteria:

* Reported allergy to egg proteins, chicken proteins, or any other constituent of the vaccine.
* Documented history of influenza infection.
* An acute illness with or without fever (temperature ≥ 100.4 °F, rectal) in the 72 hours preceding enrollment in the trial (Enrollment may be deferred).
* Clinically significant findings in vital signs or review of systems (investigator judgment; defer or exclude).
* Participation in any other interventional clinical trial within 30 days prior to enrollment up to termination of the subject's participation in the study.
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder.
* Known Human immunodeficiency virus (HIV)-positive mother.
* Prior history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from October to December 2005
Pre-assignment Details: A total of 30 subjects that met the inclusion and exclusion criteria were enrolled and vaccinated
Groups:
- Influenza Vaccine-naive Group: Participants have never received Influenza virus vaccine. They received 0.25 mL of Fluzone® vaccine on Day 0 and Day 28, respectively.
- Influenza Vaccine-primed Group: Participants have received Influenza virus vaccine in the past. They received 0.25 mL of Fluzone® vaccine on Day 0.
Period: Overall Study
Arm/Group | Influenza Vaccine-naive Group | Influenza Vaccine-primed Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine-naive Group | Influenza Vaccine-primed Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 11.92 (6.36) | 26.43 (8.00) | 19.18 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition Antibodies Pre-vaccination and 14 Days Post-vaccination
Description: GMTs and their 95% Confidence interval are presented for each of the 3 antigens in the Fluzone® vaccine 2005-2006 Pediatric formulation.
  Post-dose 1 (Influenza vaccine Primed group); post-dose 2 (Influenza vaccine Naive group)
Time Frame: Day 14 post-vaccination
Population: Geometric Mean Titers were assessed on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza Vaccine-naive Group | Influenza Vaccine-primed Group
Number analyzed (Participants) | 13 | 14
Titer
  Flu A/New Caledonia/20/99 (H1N1) - Pre | 5.0 [5.0 to 5.0] | 8.2 [4.3 to 15.6]
  Flu A/New Caledonia/20/99 (H1N1) - Post | 187.8 [105.4 to 334.5] | 95.1 [44.0 to 205.9]
  Flu A/New York/55/2004 (H3N2) - Pre | 8.5 [4.9 to 14.7] | 32.8 [10.9 to 98.4]
  Flu A/New York/55/2004 (H3N2) - Post | 328.6 [181.2 to 596.0] | 249.8 [88.1 to 708.6]
  Flu B/Jiangsu/10/2003 - Pre | 9.2 [4.6 to 18.7] | 5.3 [4.7 to 5.8]
  Flu B/Jiangsu/10/2003 - Post | 59.7 [22.7 to 156.9] | 39.0 [17.2 to 88.7]

2. Other Pre Specified Outcome: Number of Subjects Who Had Solicited Local and Systemic Reactions Post-vaccination 1
Description: Solicited local reactions: injection site erythema, injection site swelling, injection site tenderness; Solicited systemic reactions: fever (temperature), irritability, abnormal crying, drowsiness, lost appetite, and vomiting.
Time Frame: 0 to 3 days post-vaccination 1
Population: Safety analysis post-vaccination 1 was on all enrolled and vaccinated subjects, Intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Influenza Vaccine-naive Group | Influenza Vaccine-primed Group
Number analyzed (Participants) | 15 | 15
Participants
  Any Solicited Injection Site Reaction post-dose 1 | 3 | 2
  Any injection site Tenderness | 2 | 1
  Grade 3 injection site Tenderness-reduced movement | 0 | 0
  Any injection site Erythema | 1 | 1
  Grade 3 injection site Erythema (≥ 5.0 cm) | 0 | 1
  Any injection site Swelling | 1 | 1
  Grade 3 injection site Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Systemic Reactions post-dose 1 | 10 | 5
  Any Fever (≥ 100.4°F) | 1 | 2
  Grade 3 Fever (> 103.2°F) | 0 | 0
  Any Crying abnormal | 4 | 1
  Grade 3 Crying abnormal (> 3 hours) | 0 | 0
  Any Irritability | 6 | 1
  Grade 3 Irritability (Inconsolable) | 0 | 0
  Any Vomiting (per 24 hours) | 1 | 0
  Grade 3 Vomiting (≥ 6 episodes) | 0 | 0
  Any Drowsiness | 6 | 3
  Grade 3 Drowsiness (Sleeps most time) | 0 | 0
  Any Appetite lost | 4 | 1
  Grade 3 Appetite lost (Refuse most feeds) | 0 | 0

3. Other Pre Specified Outcome: Number of Subjects Who Had Solicited Local and Systemic Reactions Post-vaccination 2
Description: Solicited local reactions: injection site erythema, injection site swelling, injection site tenderness; Solicited systemic reactions: fever (temperature), irritability, abnormal crying, drowsiness, lost appetite, and vomiting
  Note: Influenza vaccine-primed group received only dose 1
Time Frame: 0 to 3 days post-vaccination 2
Population: Safety analysis post vaccination 2 was on all enrolled and vaccinated subjects, Intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Influenza Vaccine-naive Group | Influenza Vaccine-primed Group
Number analyzed (Participants) | 15 | 0
Participants
  Any solicited injection site reaction post-dose 2 | 2 |
  Any injection site Tenderness | 1 |
  Grade 3 injection site Tenderness-reduced movement | 0 |
  Any injection site Erythema | 0 |
  Grade 3 injection site Erythema (≥ 5.0 cm) | 0 |
  Any injection site Swelling | 1 |
  Grade 3 injection site Swelling (≥ 5.0 cm) | 0 |
  Any solicited systemic reactions post-dose 2 | 8 |
  Any Fever (≥ 100.4 ºF) | 5 |
  Grade 3 Fever (> 103.2 ºF) | 0 |
  Any Crying abnormal | 3 |
  Grade 3 Crying abnormal (> 3 hours) | 1 |
  Any Irritability | 5 |
  Grade 3 Irritability (inconsolable) | 0 |
  Any Vomiting (per 24 hours) | 0 |
  Grade 3 Vomiting (≥ 6 episodes) | 0 |
  Any Drowsiness | 2 |
  Grade 3 Drowsiness (sleeping most time) | 0 |
  Any Appetite lost | 3 |
  Grade 3 Appetite lost (refuses most feeds) | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from day of vaccination for 2 weeks (Influenza vaccine-Primed) and 6 weeks (Influenza vaccine naive) participants.
Arm/Group | Influenza Vaccine-naive Group | Influenza Vaccine-primed Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 13/15 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine-naive Group (N=15) | Influenza Vaccine-primed Group (N=15)
Injection site tenderness (General disorders) | 3 | 1
Injection site erythema (General disorders) | 1 | 1
Injection site swelling (General disorders) | 1 | 1
Pyrexia (General disorders) | 6 | 2
Crying (Psychiatric disorders) | 5 | 1
Irritability (Psychiatric disorders) | 8 | 1
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 6 | 3
Anorexia (Metabolism and nutrition disorders) | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Otitis media (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.